CLINICAL TRIAL: NCT04599023
Title: Assessing the Feasibility of the Multiple Sclerosis Performance Test (MSPT) Device in Routine Clinical Practice in the Swiss Healthcare System
Brief Title: Assessing the Feasibility of the MSPT Device in Routine Clinical Practice in the Swiss Healthcare System
Acronym: MSPT
Status: Terminated | Type: Observational
Why Stopped: Decision of company to no longer develop the device.
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: CH-MSG-11563
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: MS; CIS; MSFC; Contrast Sensitivity Test; Walking Speed Test; 25 foot walk; Manual Dexterity Test; Processing Speed Test; self-administrating; medical device
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MS patients including CIS: Patients with a diagnosis of MS, including Clinically Isolated Syndrome (CIS), who have the ability to understand the audio and visual instructions for the MSPT modules and whose visual function that does not preclude an ability to see the screen of the MSPT tool.
  Interventions: Device: MSPT

INTERVENTIONS:
Device: MSPT — The MS Performance Test (MSPT) software tool and accompanied hardware is an iPad®-based assessment tool, developed via collaboration between Biogen and the Cleveland Clinic Mellen Center, and designed to objectively quantify the major motor, visual and cognitive function data, and quality of life outcomes, associated with MS and related disorders.These assessment modules of the MSPT are self-administered by MS patients at the point of care and incorporate and expand upon previously validated measures of the MSFC.

SUMMARY:
The Multiple Sclerosis Functional Composite (MSFC), a reliable and well-validated instrument, was developed as a multidimensional quantitative measure of neurologic disability in MS. However, the traditional form of the MSFC has various limitations, including the need for MS patients to be assessed in a clinical setting by trained technicians, which requires additional human resources and time in a clinical routine practice setting. Furthermore, storage of MSFC data for longitudinal comparison is difficult and time consuming. The MS Performance Test (MSPT) software tool is designed to objectively quantify the major motor, visual and cognitive function data, and quality of life outcomes, associated with MS and related disorders.

This is a single center observational study that will examine the use of the MSPT in a real world setting. Study enrollment will occur at one center in Switzerland.

DETAILED DESCRIPTION:
Study participation will be offered to MS patients either on day of clinic visit. Patient screening, consent discussion and MSPT test completion is estimated to take approximately an hour prior to the appointment with the treating physician. Participants begin with an instructional overview, which acquaints them with all elements of the MSPT. The tests will be performed in the same order and if a study participant elects to discontinue testing or skip a module, they will be asked to indicate the reasons on the screen. Each module has accompanying instructions.

Upon completion of testing at first and last study visit, patients, research nurse/coordinator and treating physician will be asked to fill in a short satisfaction questionnaire related to the functionality of the MSPT.

HCPs will have the ability to view de-identified longitudinal MSPT outcomes for each patient on the MSPT tool.

De-identified data abstracted from each site will be stored in a cloud-based data repository. Access to the MSPT Cloud and data therein is restricted to the healthcare institution using the registered MSPT tool. The site will periodically send de-identified and encrypted aggregate data to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Diagnosis of MS, including Clinically Isolated Syndrome (CIS)
* Ability to understand the audio and visual instructions for the test modules
* Visual function, based on the investigator's clinical judgement, that does not preclude an ability to interact with the MSPT.

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Patients under 18 years of age will be excluded.
* Other unspecified reasons that, in the opinion of the Sponsor-Investigator, make the patient unsuitable for participation in the demonstration project. A patient only needs to complete the assessments deemed appropriate by the Sponsor-Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of MS, including Clinically Isolated Syndrome (CIS)
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who complete all modules | 2 years
  Percentage of patients who complete all modules (out of those who initiate testing) will be measured to evaluate the feasibility of the MSPT in a clinical care setting when used by MS patients.
Percentage of patients who complete each module | 2 years
  Percentage of patients who complete each module (out of those who initiate each module) will be measured to evaluate the feasibility of the MSPT in a clinical care setting when used by MS patients.
Percentage of patients who skip modules | 2 years
  Percentage of patients who skip modules (out of those who initiate testing) will be measured to evaluate the feasibility of the MSPT in a clinical care setting when used by MS patients.
Time to complete the MSPT | 2 years
  Time to complete the MSPT will be measured to evaluate the feasibility of the MSPT in a clinical care setting when used by MS patients.
Time to complete the individual MSPT modules | 2 years
  Time to complete the individual MSPT modules will be measured to evaluate the feasibility of the MSPT in a clinical care setting when used by MS patients.
Frequency of reasons for not completing test modules | 2 years
  Frequency of reasons for not completing test modules will be measured to evaluate the feasibility of the MSPT in a clinical care setting when used by MS patients.
Frequency distribution of demographic characteristics of patients who fail to complete specific MSPT modules | 2 years
  Frequency distribution of demographic characteristics (as captured in the MyHealth module) of patients who fail to complete specific MSPT modules will be measured to evaluate the feasibility of the MSPT in a clinical care setting when used by MS patients.

SECONDARY OUTCOMES:
Net promoter score based on satisfaction questionnaires | 2 years
  Net promoter score based on satisfaction questionnaires conducted with patients to probe about experience interfacing the MSPT
Net promoter score based on patient questionnaire | 2 years
  Net promoter score based on patient questionnaire related to perceived benefit of the MSPT for improved monitoring of MS disease progression
Net promoter score based on treating physician and administrator questionnaire for improved monitoring of MS disease progression | 2 years
  Net promoter score based on treating physician and administrator questionnaire related to perceived benefit of the MSPT for improved monitoring of MS disease progression
Net promoter score based on satisfaction questionnaires conducted with treating physicians and the MSPT administrator to probe about experience | 2 years
  Net promoter score based on satisfaction questionnaires conducted with treating physicians and the MSPT administrator to probe about experience interfacing the MSPT
Change in MSPT outcomes in patient subgroups of interest at baseline and at each visit over time | 2 years
  Change in MSPT outcomes in patient subgroups of interest at baseline and at each visit over time (e.g., newly diagnosed, untreated RRMS, patients with cognitive impairment, patients with cognitive impairment but only mild physical disability, patients of different area of origin)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hoepner, PD Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital Bern, Ambulantes Neurozentrum, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No